CLINICAL TRIAL: NCT05313074
Title: SARS-CoV-2 Specific Immune Response After COVID-19 Vaccination in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Thailand (Other Government)
Collaborators: Mahidol University (Other)
Responsible Party: Principal Investigator, Thanarath Imsuwansri, MD, Head of Research Division, National Cancer Institute, Thailand
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 013_2021RC_IN695
Record Dates: First submitted 2022-04-04; First posted 2022-04-06 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: COVID-19; Cancer
Keywords: COVID-19; Cancer; Immune response
MeSH Terms: conditions — COVID-19; Neoplasms | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Cancer patients and healthy volunteers will be compared for effectiveness of CoronaVac vaccine in parallel after 2 doses of vaccination for 15 days by neutralizing antibody test
Masking Description: All participants, including patients with solid tumor and healthy volunteers will be received 2 doses of CoronaVac at National Cancer Institute of Thailand between 2020-2021. Blood samples will be collected after second dose of Sinovac for 15 days and the neutralizing antibody (NAb) titers will be detected using live-virus neutralization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteers (Placebo Comparator): Healthcare workers at National Cancer Institute
  Interventions: Biological: CoronaVac vaccine
- Cancer patients (Active Comparator): Cancer patients were divided into 3 groups based on treatment status including
  1. active cancer on treatment
  2. Planned to start treatment
  3. Post-treatment (<6 months)
  Interventions: Biological: CoronaVac vaccine

INTERVENTIONS:
Biological: CoronaVac vaccine — An inactivated virus COVID-19 vaccine developed by the Chinese company Sinovac Biotech.
  Other Names: Sinovac

SUMMARY:
Our study highlights a low degree of neutralization-afforded protection mounted by CoronaVac in cancer patients when compared with healthy volunteers, especially patients who received chemotherapy. Further booster doses, beyond the conventional two-dose regimen might be needed for recipients of CoronaVac to maintain a long-term anamnestic response.

DETAILED DESCRIPTION:
A total of 311 participants, including 107 patients with solid tumor and 204 healthy volunteers who received 2 doses of CoronaVac were recruited from National Cancer Institute of Thailand between 2020-2021. Blood samples were collected after second dose of CoronaVac for 15 days and the neutralizing antibody (NAb) titers were detected using live-virus neutralization.SARS-CoV-2 antibody positivity was detected in 77 (72%) patients and 199 (97.5%) healthy volunteers. Antibody positivity rate was lowest (67.2%) in patients who received chemotherapy, followed by patients with post-treatment (74.2%) and patients who planned to start treatment (91.7%). Our study highlights a low degree of neutralization-afforded protection mounted by CoronaVac in cancer patients when compared with healthy volunteers, especially patients who received chemotherapy. Further booster doses, heterologous or otherwise, beyond the conventional two-dose regimen might be needed for recipients of CoronaVac to maintain a long-term anamnestic response.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age at least 18 years
* Patients with a diagnosis of solid tumors
* Ability to understand the patient information and study consent. Signed and dated written informed consent must be available before performing any study-related procedure
* Willing and able to comply with the study procedures.
* Willing to receive a Coronavac vaccine (Sinovac).

Exclusion Criteria:

* Patients who cannot provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Immune response of Coronavac vaccine in Thai cancer patients | 15 days after 2 doses of vaccination
  Immune response of of the inactivated COVID-19 vaccine (Coronavac) in Thai cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Thanarath Imsuwansri, MD, Principal Investigator — National Cancer Institute of Thailand
Locations (1):
- National Cancer Institute, Ratchathewi, Bangkok, Thailand